CLINICAL TRIAL: NCT00340795
Title: Media-Smart Youth Program Evaluation Study
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905197; 05-CH-N197
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-03-07

CONDITIONS: Adolescent
Keywords: Media Analysis; Nutrition; Physical Activity; After-School; Exercise
MeSH Terms: conditions — Motor Activity

SUMMARY:
This study will evaluate the impact of a Media-Smart Youth (MSY) curriculum on adolescent knowledge and behavioral intent regarding media messages, nutrition, and physical activity. The study is part of the U.S. Government's efforts to fight obesity and increase physical activity among American youth. The MSY program seeks to empower adolescents to make healthful choices about nutrition and physical activity by helping them understand how media can influence their lives. This is important because it is estimated that young people view as many as 40,000 commercial messages a year on television alone, many of which promote unhealthy snack foods and beverages.

Youth between 11 and 13 years of age who are participating in selected after-school programs in the Washington, D.C., metropolitan area may be eligible for this study.

Participants are randomly assigned to either receive the MSY curriculum or serve as controls. Youth in the MSY group participate in a workshop consisting of 10 lessons and a creative project to create a media message for their peers on the topic of nutrition and physical activity. During the sessions, the young people receive information on nutrition and physical activity and learn about media production and how to critically examine the media. Youth in the control group participate in after-school programs unrelated to MSY. All participants fill out questionnaires measuring their knowledge, skills, and behavioral intent related to media analysis, nutrition and physical activity both at the start of the study and at its completion.

DETAILED DESCRIPTION:
A. Objectives of Study

The purpose of this study is to determine the impact of the Media-Smart Youth (MSY) curriculum on adolescent knowledge skills and behavioral intent in the areas of media analysis, nutrition, and physical activity. The study asks whether youth participating in the MSY curriculum 1) increase their skills in analyzing media messages; 2) increase their knowledge of the basic principles of healthful and nutritious foods and increase their skills and behavioral intent to make healthful food choices in real-life settings; and 3) increase their knowledge of the importance of daily physical activity in promoting health and increase their skills and behavioral intent to be more active in their daily lives.

B. Study Design

The evaluation will use a group randomization design, in which 18 after-school programs will be randomly assigned to either receive the MSY curriculum or serve as controls. Nine youth-serving agencies running pre-existing structured after-school programs in the Washington, DC metropolitan area will be solicited to participate in the evaluation. For each agency, two program sites will be selected with each pair of sites matched for socioeconomic status, race and ethnicity, all factors that may affect the program outcomes. The sites will then be randomly assigned to either the treatment or control group. During the implementation of the MSY curriculum at the treatment sites, participants in the control sites will receive after-school programming unrelated to MSY. Fifteen youth in each after-school program, or 270 youth, will be recruited to participate in the study. Parental consent and youth assent will be obtained. At the end of the program implementation, program staff from the treatment and control sites will be offered training in implementing the MSY curriculum.

C. Outcome Measures

The MSY program outcomes on knowledge, skills and behavioral intent related to media analysis, nutrition, and physical activity will be measured using a paper-and-pencil self-administered questionnaire (SAQ). All 270 youth will complete the SAQ pretest before the start of the MSY curriculum. Following the completion of the curriculum, all 270 youth will complete the SAQ posttest. For the treatment of after-school participants, data collection is incorporated into the MSY curriculum delivery. Following implementation of the MSY curriculum, the treatment group facilitators will be interviewed to identify any modifications made to the ascribed curriculum. Program directors of the control groups will also be interviewed to determine the general content of the program(s) in which the control youth participated.

ELIGIBILITY:
* INCLUSION CRITERIA:

Youth aged 11-13 are the primary participants in this study.

All youth identified in either the treatment or control groups will be

included in the study.

At no point during the program implementation, including the data

collection, will any participant be excluded from the group

membership or activities.

EXCLUSION CRITERIA:

Treatment subjects who have participated in less than seven lessons will be excluded from the treatment group for the purpose of analyzing program effects.

They will, however, be included in intent-to-treat analyses to check for biases from excluding these participants.

Ages: 11 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0
Dates: Start 2005-08-04; Study Completion 2007-03-07

CONTACTS AND LOCATIONS:
Locations (1):
- Academy for Education Development, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Murray DM, Hannan PJ, Wolfinger RD, Baker WL, Dwyer JH. Analysis of data from group-randomized trials with repeat observations on the same groups. Stat Med. 1998 Jul 30;17(14):1581-600. doi: 10.1002/(sici)1097-0258(19980730)17:143.0.co;2-n. PMID 9699231